CLINICAL TRIAL: NCT04880057
Title: Effects of Agility Training on Executive Function, Dual Task Performance and Brain Activation in Healthy Adults
Brief Title: Agility Training on Executive Function, Dual Task Performance and Brain Activation in Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202103055RINB
Record Dates: First submitted 2021-05-03; First posted 2021-05-10 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Agility Training; Executive Function
Keywords: brain activity; motor performance; dual task walking; executive function; agility training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance+Aerobic training group (Active Comparator): Resistance+Aerobic training group (RAeT) RAeT includes resistance training (RT) program and aerobic training (AeT) program.
  Interventions: Other: Resistance+Aerobic training
- Agility training group (Experimental): Agility training
  Interventions: Other: Agility training

INTERVENTIONS:
Other: Resistance+Aerobic training — The RT focuses on lower extremity workout, including leg press, hamstring curls, and calf raises. The participants start with intensity at 12 RM and finished with intensity at 8 RM after 3 weeks. There are 8 repetitions, 2 sets for each action. It will take 15 minutes to complete RT.
  The AeT is composed by cycling on stationary bikes in the first week, stepping on steppers in 2nd week, and running on treadmills in the last week. Participants are asked to wear a portable heart rate monitor throughout the experiments. They have to maintain their heart rates in 60%-75% of predicted maximal heart rate (moderate intensity exercise), which has been shown to be benefit on cognition[3]. It took the participants 25 minutes to complete AeT.
  Other Names: RAeT
  Arms: Resistance+Aerobic training group
Other: Agility training — AT program consists of three parts: technical drills, pattern running and reactive agility training. There will be nine sessions over 3 weeks and progress the intensity, complexity or velocity every week.
  Other Names: AT
  Arms: Agility training group

SUMMARY:
This study will investigate the effect of agility training on executive function, dual task walking and brain activation in healthy adults. Participants (N=70) will be randomly assigned to resistance+aerobic training group (RAeT) or agility training group (AT). Participants in RAeT (n=35) will receive 15-minute lower extremity workout first and then 25-minute moderate intensity (60-75% predicted maximal heart rate) aerobic training. Participants in AT (n=35) will do the agility exercise program consisting of technical drills, pattern running and reactive agility training. The intervention will be twelve-time group intervention (3-5persons) in four weeks, 50 minutes per session (5-minute warmup, 40- minute main training, 5-minute cool-down). Participants will undergo three measurement time points (pre-, post-intervention and one month follow-up). Outcome measures will include executive function (N-back test, stroop test and Wisconsin card sort test), single and dual task walking performance and brain activity (fNIRS on prefrontal cortex, supplementary motor area and premotor cortex). Two-way analysis of variance (ANOVA) with Tukey post-hoc test will be used to examine the group x time interaction on three outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* (1) age between 20 to 30 years, and (2) ability to walk 20 meters independently without an assistive device.

Exclusion Criteria:

* (1) overweight (BMI>24), (2) any smoker or alcohol abusers, (3) suffering from chronic diseases that loss of control, (4) Unstable physiological conditions, such as abnormal signs like high blood pressure, headache, dyspnea, fever, etc., (5) any neuromuscular or cardiopulmonary diseases that would influent the exercise performance, and (6) suffering from diseases which exercises are their contraindications

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Executive function- N-back task (3-back) | Change from Baseline score at 3 weeks
  N-back task (3-back) is used to measure working memory
Executive function- N-back task (3-back) | Change from Baseline score at 7 weeks
  N-back task (3-back) is used to measure working memory
Executive function- Stroop test | Change from Baseline score at 3 weeks
  Stroop test is used to measure the selective attention and conflict resolution.
Executive function- Stroop test | Change from Baseline score at 7 weeks
  Stroop test is used to measure the selective attention and conflict resolution.
Executive function- Wisconsin card sort test | Change from Baseline score at 3 weeks
  Wisconsin card sort test is an easy way to assess the ability of mental set shifting.
Executive function- Wisconsin card sort test | Change from Baseline score at 7 weeks
  Wisconsin card sort test is an easy way to assess the ability of mental set shifting.
Single walking performance- Walking speed | Change from Baseline cadence at 3 weeks
  The unit is length (cm) per seconds
Single walking performance- Walking speed | Change from Baseline cadence at 7 weeks
  The unit is length (cm) per seconds
Single walking performance- Cadence | Change from Baseline cadence at 3 weeks
  The unit is steps per minutes
Single walking performance- Cadence | Change from Baseline cadence at 7 weeks
  The unit is steps per minutes
Single walking performance- Stride length | Change from Baseline cadence at 3 weeks
  The unit is cm
Single walking performance- Stride length | Change from Baseline cadence at 7 weeks
  The unit is cm
Single walking performance- Step duration | Change from Baseline cadence at 3 weeks
  The unit is seconds
Single walking performance- Step duration | Change from Baseline cadence at 7 weeks
  The unit is seconds
Dual task walking performance- Walking speed | Change from Baseline cadence at 3 weeks
  The unit is length (cm) per seconds
Dual task walking performance- Walking speed | Change from Baseline cadence at 7 weeks
  The unit is length (cm) per seconds
Dual task walking performance- Cadence | Change from Baseline cadence at 3 weeks
  The unit is steps per minutes
Dual task walking performance- Cadence | Change from Baseline cadence at 7 weeks
  The unit is steps per minutes
Dual task walking performance- Stride length | Change from Baseline cadence at 3 weeks
  The unit is cm
Dual task walking performance- Stride length | Change from Baseline cadence at 7 weeks
  The unit is cm
Dual task walking performance- Step duration | Change from Baseline cadence at 3 weeks
  The unit is seconds
Dual task walking performance- Step duration | Change from Baseline cadence at 7 weeks
  The unit is seconds
Dual task walking performance- the correct rates of arithmetic task | Change from Baseline cadence at 3 weeks
  The participants will be instructed to subtract by 7 serially from a 3-digit number while walking at their fastest speed in dual task walking condition
Dual task walking performance- the correct rates of arithmetic task | Change from Baseline cadence at 7 weeks
  The participants will be instructed to subtract by 7 serially from a 3-digit number while walking at their fastest speed in dual task walking condition

SECONDARY OUTCOMES:
Brain activities over premotor cortex- Executive function | Change from Baseline at 3 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over premotor cortex- Executive function | Change from Baseline at 7 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over supplementary motor area- Executive function | Change from Baseline at 3 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over supplementary motor area- Executive function | Change from Baseline at 7 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over primary motor cortex- Executive function | Change from Baseline at 3 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over primary motor cortex- Executive function | Change from Baseline at 7 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over premotor cortex- Single walking | Change from Baseline at 3 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over premotor cortex- Single walking | Change from Baseline at 7 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over supplementary motor area- Single walking | Change from Baseline at 3 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over supplementary motor area- Single walking | Change from Baseline at 7 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over primary motor cortex - Single walking | Change from Baseline at 3 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over primary motor cortex - Single walking | Change from Baseline at 7 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over premotor cortex- Dual task walking | Change from Baseline at 3 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over premotor cortex- Dual task walking | Change from Baseline at 7 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over supplementary motor area- Dual task walking | Change from Baseline at 3 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over supplementary motor area- Dual task walking | Change from Baseline at 7 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over primary motor cortex - Dual task walking | Change from Baseline at 3 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over primary motor cortex - Dual task walking | Change from Baseline at 7 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan